CLINICAL TRIAL: NCT04297189
Title: A Pilot Program Measuring Effectiveness of Health Coaching Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Senior Cardiologist, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HMO-0018-19
Record Dates: First submitted 2019-10-27; First posted 2020-03-05 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Sedentary Behavior; Nutritional and Metabolic Disease
MeSH Terms: conditions — Sedentary Behavior; Metabolic Diseases

STUDY DESIGN:
Masking Description: each participant will receive a coding number and the key will be kept in the primary investigator offices.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coaching Intervention (Experimental): Single arm pilot study of coaching intervention
  Interventions: Behavioral: Coaching and health information intervention

INTERVENTIONS:
Behavioral: Coaching and health information intervention — 8 session intervention with,group meetings with coaching tools and health information on nutrition and physical activity and coping with stress.

SUMMARY:
Women will participate in a workshop within a group and individual meetings. the workshop will include providing information regarding guidelines for healthy eating, engaging in physical activity, personal training tools to build self-efficacy and to encourage implementing a healthy life style.

DETAILED DESCRIPTION:
Participants are interviewed for eligibility and if appropriate sign consent and undergo measurements of weight, height and blood pressure.

At the first meeting there is a pre-study questionnaires and initial coaching session

Eight group meetings will take place and will include:

up-to-date knowledge on nutrition (by a dietitian), exercise (by a physiotherapist) and coping skills for stress (by a psychologist).

Additionally the meetings will also include coaching tools which the participants will practice during the session. The multidisciplinary team has been trained in coaching tools to evaluate in group settings.

In the last meeting, participants will be asked to fill out post study questionnaires measurements will be taken (weight and blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* over age 18
* Women who agree to fill out questionnaires
* Women who agree to attend sessions (attending 80% of sessions)
* Women who are fluent in Hebrew

Exclusion Criteria:

* Pregnancy
* Women with significant untreated psychiatric diagnosis
* Insulin-dependent diabetes
* End-stage renal disease
* Unstable Angina
* Women who are not fluent in Hebrew
* Women currently treated by multidisciplinary staff (eg, heart failure, cardio rehabilitation)
* Women who have been enrolled in other programs of the center at the discretion of the staff will not be included in the study
* Women who do not want to make a healthy lifestyle change
* Failure to reach 75% of sessions during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
self efficacy | 1 year
  Change in (improved) self efficacy as assessed by Tschannen-Moran Moore score
Behavioral change | 1 year
  achieved 80% of the goal they set in first meeting or achieved the goal 80% of the time

SECONDARY OUTCOMES:
nutrition | 1 year
  adaptation of the Israeli Ministry of Health Diet Scale
physical activity | 1 year
  increase in self-report of exercise in minutes per week
weight | 1 year
  kg
experiential avoidance | 1 year
  Reduction on experiential avoidance as measured on the Brief Experiential Avoidance Scale

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Reinfeld, RN, Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel